CLINICAL TRIAL: NCT06271486
Title: Pregabalin as Alternative to Epidural Blood Patch in Treatment of Postdural Puncture Headache: A Randomized Controlled Clinical Trial
Brief Title: Pregabalin in Treatment of Postdural Puncture Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC. 40.5.2023
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Pregabalin; Conservative Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (pregabalin group) (Active Comparator): Received oral pregabalin treatment administered at 150 mg daily, with 75 mg given every 12 hours.
  Interventions: Drug: Pregabalin 75mg
- Group B (EBP group) (Active Comparator): Received active therapy in the form of an EBP and Group C (control group) received conservative treatment.
  Interventions: Biological: An epidural blood patch (EBP)
- Group C (the control group) (Active Comparator): received conservative treatment.
  Interventions: Combination Product: conservative treatment.

INTERVENTIONS:
Drug: Pregabalin 75mg — Group A (pregabalin group) received oral pregabalin treatment administered at 150 mg daily, with 75 mg given every 12 hours.
  Arms: Group A (pregabalin group)
Biological: An epidural blood patch (EBP) — Group B (EBP group) received active therapy in the form of an EBP
  Arms: Group B (EBP group)
Combination Product: conservative treatment. — Group C (control group) received conservative treatment providing recommendations to the patients, including 24 hours of bed rest, stool softener, and consuming a minimum of 2.0 liters of fluid daily. Analgesics were permitted for pain relief depending on the patient's disease status.
  Arms: Group C (the control group)

SUMMARY:
Lumbar puncture (LP), often known as a "spinal tap," is a standard medical technique pioneered in the late 1900s by Heinrich Quincke. It involves the retrieval and analysis of cerebrospinal fluid (CSF) from the spinal cord, serving as the benchmark for diagnosing conditions like subarachnoid hemorrhage, meningitis, and specific neurological conditions. Pregabalin, an anticonvulsant medicine that blocks calcium entry, is used to treat a variety of diseases. It has been used to relieve pain in a variety of patient groups, including those with chronic pain, epilepsy, and anxiety disorders

ELIGIBILITY:
Inclusion Criteria:

* age from 21 to 65 years old,
* both genders,
* confirmed diagnosis of postdural puncture headache (PDPH)

Exclusion Criteria:

* patient refusal
* known allergy to the drug used in the study
* patients with a history of convulsions
* chronic headaches
* contraindications to regional anesthesia (such as local infection and coagulation abnormalities).
* Clinical indications of elevated intracranial pressure or associated risk factors
* Deteriorated patients

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
the incidence of complete relief | 48 hours
  The incidence of complete relief, as reflected in the success rate of the intervention at 48 hours.

SECONDARY OUTCOMES:
The intensity of the headache | 48 hours
  The intensity of the headache was measured using visual analogue score (VAS). The scale uses a scoring system in which values of 0, 1-3, 4-6, and 7-10 correspond, respectively, to the absence of pain, mild, moderate, and severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Neveen Kohaf, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request from corresponding author
Supporting Information: Study Protocol, SAP, ICF